CLINICAL TRIAL: NCT03078387
Title: Bilateral Retinal Embolic Phenomena Always Necessitates Immediate and Intensive Investigation. Careful, Documented, Ophthalmic Examination is All we Require to Initiate Life Saving Investigations.
Brief Title: The Extreme Significance of Bilateral Embolic Retinal Phenomena That Can be Life Saving
Status: Completed | Type: Observational
Sponsor: Dr. Shawkat Michel (Other)
Responsible Party: Sponsor-Investigator, Dr. Shawkat Michel, Principal Investigator, Dr. S.S. Michel Clinic
Organization: Dr. S.S. Michel Clinic (Other)
Other Study IDs: Bilateral retinal emboli
Record Dates: First submitted 2017-03-06; First posted 2017-03-13 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Life Threatening Diseases; Embolic Shower
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: imaging — imaging before and after treatment
  Other Names: color fundus photos

SUMMARY:
This study shows how careful ophthalmic examination of two patients showed signs of simultaneous bilateral retinal emboli. Starting from this point significant, life threatening, underlying reasons were found and treated.

DETAILED DESCRIPTION:
Two patients were found to have signs of simultaneous bilateral retinal emboli. One patient was asymptomatic and routine ophthalmic examination showed bilateral retinal hemorrhages and exudates close to both optic discs. This patient was on anti-coagulant treatment for atrial fibrillation. The finding of bilateral signs of retinal emboli necessitated immediate blood tests and dose adjustments of her medication.

The second case did not have general symptoms other than mild evening chills and her eye examination again was the start point of intensive investigation to find the reason of her bilateral retinal emboli. Ultrasound studies revealed a life threatening reason that was urgently treated.

ELIGIBILITY:
Inclusion Criteria:

* any patient who is found to have sure signs of bilateral retinal emboli.

Exclusion Criteria:

* all other bilateral retinal diseases.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any patient in which signs of bilateral retinal emboli are seen and documented (imaged).
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2006-08-31 (Actual); Primary Completion 2013-01-29 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The extreme significance of immediate investigation of cases of bilateral retinal emboli (non-diabetic bilateral posterior pole retinal nerve fiber or pre-retinal hemorrhages). | through study completion, an average of one year
  Patients that are noticed to have signs of bilateral retinal emboli (bilateral retinal nerve fiber layer hemorrhages or bilateral pre-retinal hemorrhages and sometimes bilateral soft exudates) may be asymptomatic or have very mild symptoms. However these patients must be immediately and, if needed, intensively investigated to find the source of these emboli. The extremely important point of this study is these patients usually have life threatening conditions that should be found out and treated in time.

CONTACTS AND LOCATIONS:
Overall Officials: shawkat s. Michel, MD, FRCS Ed, Principal Investigator — Dr. S.S. Michel Clinic, 214 MHC, 156 street and 87 Ave, Edmonton, AB, Canada
Locations (1):
- Dr. S.S. Michel Clinic, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Color photographs of patients with bilateral retinal emboli and relevant medical conditions will be shared.
Time Frame: Color photographs are available from the time of publishing and until the end of 2018.
Access Criteria: Ophthalmologists interested may request the color photos by mail or email. Within four weeks from receiving request color photos will be sent